CLINICAL TRIAL: NCT02686307
Title: Predicting Blood Pressure in Patients Following Defibrillation in Patients With an ICD Implant
Brief Title: Predicting Blood Pressure in Patients Following Defibrillation
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 00013500
Record Dates: First submitted 2007-12-21; First posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Blood Pressure
MeSH Terms: interventions — Defibrillators, Implantable

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICD Implant: All patients receiving a dual chamber ICD
  Interventions: Procedure: ICD Implant

INTERVENTIONS:
Procedure: ICD Implant — Implantation of an implantable cardioverter/defibrillator
  Other Names: implantable cardioverter defibrillator; Medtronic; St Jude Medical; Boston Scientific

SUMMARY:
During tachyarrhythmias, central venous pressures increases while arterial blood pressure (BP) decreases. The result is mixed messages to the central nervous system. On one hand, the unloading of the arterial baroreceptors results in reflex tachycardia and an increase in sympathetic nerve activity (SNA). On the other hand, the increase in filling pressure and thus the activation of the cardiopulmonary baroreceptors result in reflex bradycardia and sympathoinhibition. The investigators have previously shown that during supraventricular and ventricular tachycardia, arterial baroreflex gain (BRG) predominates with minimal contribution from the cardiopulmonary BRG. In addition, the investigators found that arterial BRG directly correlates with BP recovery following tachycardia termination. The roles of the arterial and cardiopulmonary BRGs during ventricular fibrillation (VF) however, remain unknown. Furthermore, the role of the arterial BRG in determining 1) BP recovery following VF induction and 2) the frequency of ventricular tachycardia (VT)/VF events in patients undergoing implantation of an implantable cardioverter/defibrillator (ICD) remain unknown. Analysis of the changes in sinus node cycle length during VF inductions in patients undergoing the implantation of a dual chamber or triple chamber ICD, provide a unique opportunity at looking at the autonomic changes that accompany VF.

DETAILED DESCRIPTION:
Design: This is a prospective, non-randomized study. The purpose of the present study is 1) to assess whether the changes in sinus node cycle length during VF induction following ICD implant correlate with arterial BRG, and 2) to determine whether these changes, and thus arterial BRG, predict BP recovery post-defibrillation.

POSSIBLE BENEFITS: There are no specific potential benefits for subjects participating in this study. Results from this study should greatly improve investigator's knowledge of VF and BP control.

POSSIBLE RISKS & DISCOMFORTS: The potential risks or discomforts are associated with the assessment of arterial baroreflex gain.

Nitroprusside (NTP) infusion may result in significant drop in blood pressure, heart attack, rhythm disturbances and stroke. The risks associated with phenylephrine (PE) infusion include blood pressure elevation, heart attack, rhythm disturbances and stroke. The likelihood of this is very small since the medications will be given in small, gradual doses with close monitoring by study personnel and physicians. If significant blood pressure changes occur, the medication will be stopped immediately. Stopping the medication will quickly reverse any blood pressure changes since the drugs have a very short half-life.

Study procedures: Arterial baroreflex gain measurements will be performed either at the patient's bedside or in the electrophysiology laboratory as described below. BP will be monitored using a non-invasive arterial tonometer (Colin, San Antonio, TX) if performed at bedside, or a preexisting arterial line if performed in the laboratory. Logistical considerations, such as timing, would be a reason for performing the assessment at the bedside. The majority of the studies will be performed in the laboratory. This procedure will take approximately 20 minutes.

NTP will be injected into a peripheral vein as bolus infusion starting with 50mcg and increasing in 50mcg increments. NTP administration will be stopped when a 20-30mmHg drop in systolic or diastolic blood pressure is elicited. This will be followed by PE administration as a bolus infusion starting with 50mcg and increasing in 50mcg increments. PE administration will be stopped when an increase in systolic or diastolic BP of 10-20 mmHg above baseline is elicited. If, at any time during drug infusion, systolic blood pressure decreases below 90mmHg or increases above 160mmHg, or if the subject complains of discomfort that could be associated with blood pressure changes, the infusion will stop immediately. Specific conditions will result in arterial BRG being assessed using only NTP or PE: 1) allergy to NTP, or a systolic blood pressure (SBP) <100 will exclude the use of NTP; 2) hypersensitivity to phenylephrine products, narrow angle glaucoma or a SBP >140mmHg will exclude the use of PE. Drugs will be infused through existing venous access.

Arterial BRG will be determined as change in heart rate (HR)/change in diastolic blood pressure (DBP) during drug infusion.

Following assessment of baroreflex gain, (patients will be moved to the laboratory if the assessment was performed at bedside) patients will undergo their scheduled procedure. After the implantation of their ICD, VF induction is performed for the assessment of the defibrillation thresholds.

During the VF episodes, changes in sinus node CL measured from the stored atrial electrogram (EGM) from the implanted device will be recorded. Specifically, investigators will be measuring the average CL over the last 5 seconds before defibrillation (VF-SNCL) and will be comparing it with the average sinus node CL during the 5 seconds prior to VF induction (Baseline-SNCL). In addition, continuous BP monitoring from an existing arterial line during and following defibrillation will be stored onto a data recording system. BP recovery will be defined as the difference in mean BP during the 5 seconds before defibrillation compared with the first 30 seconds after successful defibrillation. Post-shock pacing will always be set at 40bpm in a VVI mode.

The changes in sinus node CL and BP recovery measurements will only be derived from the first successful VF induction followed by successful VF termination. The induction of non-sustained VF or VT will be considered grounds for withdrawal. On the other hand, the failure to induce VF will not be considered grounds for withdrawal.

12 Month Follow-Up: Data will be gathered from scheduled and unscheduled ICD related hospital visits for 12 months. All ICD related events will be monitored and recorded. Appropriate ICD events will be defined as all events that required anti-tachycardia pacing (ATP) or defibrillation, and which were diagnosed by 2 independent electrophysiologists as being ventricular in origin.

ELIGIBILITY:
Inclusion Criteria:

1. Indication for the implantation of an ICD with atrial lead placement
2. Presence of normal sinus rhythm
3. Age 18 or older

Exclusion Criteria:

1. Moderate to severe aortic stenosis
2. Embolic stroke within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2005-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Correlation of sinus node cycle length to arterial baroreflex gain | up to 12 months
  Assessment of whether changes in sinus node cycle length during ventricular fibrillation induction correlate with arterial baroreflex gain at scheduled and unscheduled implantable cardioverter/defibrillator related hospital visits for up to 12 months

SECONDARY OUTCOMES:
Blood pressure recovery post-defibrillation | first 30 seconds after successful defibrillation
Frequency of tachyarrhythmic events | 6 months following ICD implant

CONTACTS AND LOCATIONS:
Overall Officials: Mohomed Hamdan, MD, Principal Investigator — University of Utah

IPD SHARING:
Plan to Share IPD: No